CLINICAL TRIAL: NCT07349459
Title: Clinical Study Evaluating Cardioprotective Effect of Melatonin Versus Vitamin D in Breast Cancer Patients Receiving Doxorubicin
Brief Title: Cardioprotective Effect of Melatonin Versus Vitamin D in Breast Cancer Patients Receiving Doxorubicin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Majed Essa Alharbi, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36265MD408/5/25
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-04

CONDITIONS: Melatonin; Breast Cancer Patients Diagnosed; Vitamin D Concentration; Doxorubicin
Keywords: Vitamin D; Doxorubicin; Cardioprotective Effect; Melatonin; Breast Cancer Patients

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Doxorubicin group) (Placebo Comparator): 30 patients will receive a traditional chemotherapeutic agent (Doxorubicin group) for 12 weeks.
  Interventions: Drug: Group 1 (Doxorubicin group)
- Group 2 (Vitamin D group) (Experimental): patients with Vitamin D supplementation (1000 iu/day) plus Doxorubicin for 12 weeks
  Interventions: Drug: Group 2: Vitamin D group
- Group 3 (melatonin group) (Experimental): 30 patients with 10 mg of melatonin orally, once daily plus Doxorubicin for 12 weeks.
  Interventions: Drug: Group 3: melatonin group

INTERVENTIONS:
Drug: Group 1 (Doxorubicin group) — 30 patients will receive a traditional chemotherapeutic agent (Doxorubicin group) for 12 weeks.
  Arms: Group 1 (Doxorubicin group)
Drug: Group 2: Vitamin D group — patients with Vitamin D supplementation (1000 iu/day) plus traditional therapy for 12 weeks
  Arms: Group 2 (Vitamin D group)
Drug: Group 3: melatonin group — patients with 10 mg of melatonin orally, once daily plus traditional therapy for 12 weeks
  Arms: Group 3 (melatonin group)

SUMMARY:
This study aims to assess the cardioprotective effect of melatonin and vitamin D in breast cancer patients who receive doxorubicin.

DETAILED DESCRIPTION:
Doxorubicin is one of the most potent chemotherapeutic agents and is widely used for the treatment of various cancers and hematological malignancies . Although Doxorubicin has a potential beneficial effect in cancer treatment, its dose-dependent cardio toxicity is considered a major challenge.

Doxorubicin is known to generate free radicals either by redox cycling between a semiquinone form and a quinone form or by forming a Doxorubicin-Fe3+ complex . In both pathways, molecular oxygen is reduced to superoxide ion , which is converted to other forms of reactive oxygen species such as hydrogen peroxide and hydroxyl radical . These free radicals could then cause membrane and macromolecule damage, both of which lead to injury to the heart, an organ that has a relatively low level of antioxidant enzymes such as superoxide dismutase and catalase .

Furthermore, it was revealed that Doxorubicin may enhance the death of cardiomyocytes by affecting the tumor necrosis factor signaling pathway via increasing the expression and levels of inflammatory genes interleukin and interleukin -6 .

To alleviate DOX-induced toxicity, researchers have tested a number of strategies, including the administration of antioxidants and/or antiapoptotic agents, in both in vitro and in vivo models of Doxorubicin induced cytotoxicity, but most of these trials have failed to translate into clinical benefits . As a result, there are no effective approaches for alleviating Doxorubicin induced cytotoxicity despite intensive research over recent decades .

Melatonin is a natural hormone that is primarily secreted by the pineal gland and functions as a major regulator of circadian rhythms in humans . Melatonin also plays a variety of biological roles as a modulator of mood, sexual behavior and sleep; low levels or a deficiency of melatonin are also associated with Parkinson's disease, Alzheimer's disease, epilepsy, ischemic injury, diabetes, and even cancer .

Melatonin has emerged as a promising adjuvant that protects against doxorubicin-induced cytotoxicity, as highlighted by various studies and clinical trials that have demonstrated cardioprotective effects against several chemotherapeutic agents . Moreover, melatonin exhibits low toxicity and easily enters cells owing to its good solubility in both aqueous and organic phases and its highly lipophilic properties . Vitamin D plays an important role in the regulation of body function including the cardiovascular system .

Vitamin D deficiency results in the decrease of active calcitriol leading to inhibition of proliferation of cardiomyocytes and vascular smooth muscles .

This study aims to assess the cardioprotective effect of melatonin and vitamin D in breast cancer patients who receive doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old.
* Gender: female.
* Positive breast cancer women who are scheduled to receive Doxorubicin.
* Have a good performance status according to the eastern cooperative oncology group with a score of 0-2.
* Normal baseline Echocardiography with left ventricular ejection fraction ≥ 50%.
* Normal renal and liver function tests.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Women with HER-2 positive of breast cancer.
* Formerly treated with Doxorubicin.
* Patients with a known hypersensitivity to any of the used drugs.
* On other concomitant vitamins or food supplements.
* Valvular heart disease, coronary artery disease, history of congestive heart failure or cardiomyopathy.
* Impaired Left ventricular systolic function in which the Left Ventricular Ejection Fraction < 50%.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Decreasing incidence and severity of cardiotoxicity | 12 weeks
  Assessment of decreasing incidence and severity of cardiotoxicity by echocardiogram and ejection fraction is associated with doxorubicin treatment.

SECONDARY OUTCOMES:
change in the serum level of the (biological markers). | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be available when needed
Supporting Information: Study Protocol, ICF